CLINICAL TRIAL: NCT03720002
Title: HF2 Therapy in the Treatment of Active Ulcerative Colitis:
Brief Title: HF2 Therapy in the Treatment of Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-17-4232-UK-CTIL
Record Dates: First submitted 2018-10-21; First posted 2018-10-25 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2021-11

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: After an initial open-label run-in (if successful) the patients will be randomized to receive HF2 or placebo (2:1 allocation)
Who Masked: Participant, Care Provider, Investigator
Masking Description: participant/care provider/investigator blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental): Will receive HF2 add-on
  Interventions: Dietary Supplement: HF2
- Placebo (Placebo Comparator): Will receive placebo
  Interventions: Dietary Supplement: HF2

INTERVENTIONS:
Dietary Supplement: HF2 — placebo

SUMMARY:
This is a phase I-II study with the herbal formulation (HF2) for treatment of active ulcerative colitis

This will be a two-stage study:

Stage 1 will comprise an open label single arm exploratory study of 10 active ulcerative colitis (UC) patients investigating oral HF2 therapy for induction of remission in outpatients with active UC. Active disease is defined as (SCCAI) score ≥5 and a score of ≥2 in the modified Mayo endoscopic sub-score. Clinical remission is defined as a SCCAI score of ≤2 The patients will receive HF2 therapy for 4 weeks. Stage 2: If clinical response (defined as a drop of ≥3 points of the SCCAI score ) is achieved in ≥ 3 patients and no significant safety signals will emerge, the investigators will proceed to a prospective pilot randomized placebo-controlled study. Patients will be randomized into one of two arms: HF2 once daily or placebo formulation (2:1 proportion) for 8 weeks.

The primary outcome for stage 2 is a co-primary outcome of clinical response (reduction in SCCAI of ≤3 OR achievement of clinical remission defined as SCCAI ≤2) coupled with an objective evidence of response (Mayo score improvement of ≥1 or 50% FcAL reduction) at week 8.

Patients clinically responding at week 8, will be eligible to continue in an 8-weeks extension study to receive either placebo or 1.5gr/day curcumin alone until week 16, as per their original allocation. Exploratory analysis of outcomes for the extension study will include the percentage of patients in clinical remission (SCCAI≤2) and the percentage of patients who maintained clinical response (reduction in SCCAI of ≥3 point compared to week 0).

DETAILED DESCRIPTION:
1.1 Objective: To investigate the efficacy and safety of HF2 to induce remission in patients with active UC.

1.2 Methods:

This will be a two-stage study:

Stage 1 will comprise an open label single arm exploratory study of 10 active UC patients investigating HF2 therapy for induction of remission in outpatients with active UC.

Stage 2: If clinical response is achieved in ≥ 3 patients and no significant safety signals will emerge, the investigators will proceed to a prospective pilot randomized placebo-controlled study.

Stage 1: Open label study

1.7 Primary outcome stage I The primary outcome will be the percentage of patients in clinical remission (SCCAI score of ≤2) at week 4 after initiation of therapy

Secondary outcomes (phase 1):

1.7.1 The percentage of patients who had a rapid clinical response at day 7 after induction of therapy 1.7.2 The percentage of patients who had a clinical response at week 4 after initiation of therapy 1.7.3 Improvement in endoscopic score at week 4 compared to baseline according to modified endoscopic Mayo score (improvement of ≥ 1 point) 1.7.4 Achievement of mucosal healing (endoscopic modified Mayo score of ≤1). 1.7.5 Percentage of patients who achieve normalization and/or >50% improvement in C-reactive protein (CRP) and/or calprotectin levels (computed out of patients with abnormal values at baseline for these indices).

1.7.6 Time-to-response defined as number of days to achieve a drop of ≥3 points of the SCCAI score.

1.7.7. Time-to-ceasing of bleeding, defined as number of days for complete absence of blood in stools (SCCAI bleeding sub-score of 0), in those patients who has at least some blood in stool at entry (SCCAI bleeding sub-score of 1 or more).

1.7.8 The percentage of patients in clinical remission at day 7 after induction of therapy.

1.7.9. Improvement in IBD quality of life as gauged by questionnaire (IBDQ). 2 Intervention: Patients diagnosed with active UC will receive HF2 therapy for 4 weeks. 3 Procedures: 3.2 At inclusion: clinical and endoscopic assessment, blood and stool tests, cardiac echo and liver ultrasonography 3.4 clinical and endoscopic assessment, blood and stool tests, cardiac echo and liver ultrasonography

Stage II: A multicenter randomized placebo controlled trial. The study will be performed in Sheba Medical Center and up to 2 additional European centers (TBD). For this stage of the trial , the patients will received HF2 combintation or similar (as described above) (2:1 allocation) for 8 weeks. After completion of 8 weeks, all responders previously on active drug will receive additional 8 weeks of oral curcumin or placebo as per original arm.

Primary outcome: a composite outcome of clinical response (reduction in SCCAI of ≤3 OR achievement of clinical remiision defined as SCCAI ≤2) coupled with an objective evidence of response ( Mayo score improvement of ≥1 or 50% FcAL reduction ) at week 8

Secondary outcomes:

* Percentage of patients in clinical remission (SCCAI≤2) at week 8
* The percentage of patients who had a clinical response at week 8 after initiation of therapy
* Improvement in endoscopic score at week 8 compared to baseline according to endoscopic Mayo score (improvement of ≥ 1 point)
* Achievement of mucosal healing (endoscopic modified Mayo score of ≤1) at week 8
* Percentage of patients who achieve normalization and/or >50% improvement of CRP and/or calprotectin levels (computed out of patients with abnormal values at baseline for these indices) at week 8.
* Percentage of patients in corticosteroid-free clinical remission at week 8
* Improvement in IBD quality of life as gauged by questionnaire (IBDQ).
* Percentage of patients in clinical remission at week 16
* Percentage of patients with clinical response at week 16
* Percentage of patients with normalized fecal calprotectin and CRP

6.2. Intervention: Patients will be randomized into one of two arms: HF2 or placebo formulation (2:1 proportion) for 8 weeks. Following the first 8 weeks, responders w ill receive an additional 8 weeks of curcumin 1.5 g/d or placebo (as per original arm).

Patients will undergo clinical, laboratory (CRP, biomarkers, blood chemistry, CBC_biomarker (CRP and fecal calprotectin, at week 0,4,8 and 16 , and endoscopic assessment at baseline and week 8. Cardiac echo and liver US will be performed at week 0 and 8.

Corticosteroid tapering will be allowed as per treating physician's discretion after week 8.

ELIGIBILITY:
Inclusion criteria:

* Established diagnosis of UC
* Age- 18-70
* active UC defined by a Simple Clinical Colitis Activity Index (SCCAI) score ≥5 and a score of ≥2 in the modified Mayo endoscopic sub-score.
* Stable medication dose or if the patient has discontinued previous treatment :

for Infliximab or Vedolizumab - at least one month after patient received last dose; for Adalimumab, Golimumab, immunomodulator, corticosteroids, 5ASA - at least two weeks after patient received last dose.

Exclusion criteria:

* non-controlled renal or liver disease, hypertension, cardiovascular disease, cerebrovascular disease, chronic pancreatitis, diabetes mellitus, gallstone disease, uncontrolled migraines or neurological disorders
* significant laboratory abnormalities, including anemia with hemoglobin <10, leucopenia , thrombocytopenia , abnormal coagulation tests , or elevation of liver or kidney function tests above the normal values.
* active infection, sepsis or pneumonia.
* pregnancy/nursing
* known allergy to the compound

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Stage I: Clinical remission | week 4
  achievement of remission in the symptoms of the disease (defined as Simple Clinical Colitis Activity Index -SCCAI score of ≤2)

CONTACTS AND LOCATIONS:
Locations (2):
- Evaggelismos medical center, Athens, Greece
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ben-Horin S, Salomon N, Karampekos G, Viazis N, Lahat A, Ungar B, Eliakim R, Kuperstein R, Kriger-Sharabi O, Reiss-Mintz H, Yanai H, Dotan I, Zittan E, Maharshak N, Hirsch A, Weitman M, Mantzaris GJ, Kopylov U. Curcumin-QingDai Combination for Patients With Active Ulcerative Colitis: A Randomized, Double-Blinded, Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2024 Feb;22(2):347-356.e6. doi: 10.1016/j.cgh.2023.05.023. Epub 2023 Jun 9. PMID 37302449